CLINICAL TRIAL: NCT02917577
Title: A Randomized Controlled Trial of Two Hepatitis A Vaccine Doses Among Adolescents With Juvenile Idiopathic Arthritis and Crohn's Disease on Immunosuppressive Therapy: A Pilot Study
Brief Title: Hepatitis A Vaccine Dosing Regimens Among Pediatric Patients on Immunosuppressive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Heinrike Schmeling, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HEP-2016
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Autoimmune Rheumatologic Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avaxim Pediatric® (Active Comparator): 2 doses (0.5 mL each) six months apart of Avaxim Pediatric®
  Interventions: Biological: Avaxim Pediatric®
- Avaxim ® (adult) (Active Comparator): 2 doses (0.5 mL each) six months apart of Avaxim ® (adult)
  Interventions: Biological: Avaxim ® (adult)

INTERVENTIONS:
Biological: Avaxim Pediatric® — 2 doses (0.5 mL each) 6 months apart of Avaxim Pediatric® vaccine.
  Arms: Avaxim Pediatric®
Biological: Avaxim ® (adult) — 2 doses (0.5 mL each) 6 months apart of Avaxim ® (adult) vaccine.
  Arms: Avaxim ® (adult)

SUMMARY:
The study is a prospective, single centre, double-blinded randomized controlled trial whose goal is to compare the immune response of a population of immunosuppressed pediatric rheumatology patients on immunosuppressive medications to two different doses of Hepatitis A vaccine. The objectives are (a) to confirm that adolescents, like their adult counterparts, have a reduced immune response to hepatitis A vaccine, and (b) to compare the immunogenicity of two different dosing options of vaccine for this age group after one and two doses. A total of 60 adolescents aged 12 - 15 years with confirmed chronic rheumatologic conditions for which they are being treated with an immunosuppressive therapy will be recruited from the Rheumatology Clinic at Alberta Children's Hospital (ACH). Those found to have no immunity to hepatitis A will be enrolled. Informed, written consent will be obtained from the parent or guardian of subject, with assent obtained from the study subjects. Subjects will be randomly assigned to two doses of either Avaxim Pediatric® or Avaxim ® (adult) vaccine (Sanofi Pasteur Canada), six months apart, with hepatitis A titres done at baseline and one month after each dose. Both formulations are licensed for this age group.

DETAILED DESCRIPTION:
This is a prospective, single centre, randomized, controlled trial comparing immune responses to two doses of a licensed Hepatitis A vaccine in children. Subjects will receive 2 doses (0.5 mL each) of the assigned study vaccine (Avaxim Pediatric® or Avaxim ® (adult) vaccine). One lot of each vaccine formulation will be studied. All subjects will provide safety observations using a diary and sequential blood samples will be obtained to measure serologic/immunologic responses.

The study population will include 60 subjects with confirmed rheumatologic condition on immunosuppressive medication, males and females, in the age range 12 - 15 years. The maximum age at enrollment is 15 years and 5 months, to allow for up to 7 months in which to complete 2 doses of vaccine before age 16 years.Both vaccine formulations used in this trial has been licensed for use in Canada in the age range of the subjects being studied.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided for the subject by a parent or legal guardian.
* Written informed assent from the participants themselves.
* Subjects whose parents the investigator believes can and will comply with the requirements of the protocol (i.e. return for follow-up visits, record safety observations, able to converse with study personnel and contactable by telephone).
* Age 12 years to 15 years and 5 months
* Confirmed chronic rheumatologic condition
* Maintained on any immunosuppressive medication with the exception of pulse steroids

Exclusion Criteria:

* Systemic hypersensitivity to any Hepatitis A vaccine component such as neomycin, 2-phenoxyethanol, formaldehyde, aluminum hydroxide, Medium 199 Hanks, or Polysorbate 80.
* Thrombocytopenia or any bleeding disorder that contraindicates IM injection or blood collection.
* Receipt of blood or any blood-derived products (including IVIG) within the past 3 months.
* Previous laboratory-confirmed infection with Hepatitis A
* Previous vaccination with any Hepatitis A vaccine

The following conditions are temporary or self-limiting exclusions so a subject can be vaccinated once the condition has resolved and no other exclusion criteria exist:

* Current febrile illness or oral temperature of ≥ 38.5 °C (or equivalent by other route) or other moderate to severe illness within 24 hours before study vaccine administration
* Receipt of any Hepatitis B vaccine within 28 days of planned study vaccine doses. When Twinrix® has been studied, the response to Hepatitis B is amplified by the presence of Hepatitis A. It is unknown whether the reverse is also true.
* Routine childhood vaccines (except MMR and Varicella) must be separated from a study vaccination by at least 7 days.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinrike Schmeling, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital/University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avaxim Pediatric® | Avaxim ® (Adult)
Started | 10 | 9
Completed | 9 | 7
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avaxim Pediatric® | Avaxim ® (Adult) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 19
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 5 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 9 | 19
Diagnosis [Number; unit: participants]
  JIA | 9 | 7 | 16
  Crohn | 1 | 2 | 3
Conventional and Biologic Disease Modifying Anti-Rheumatic Drugs [Number; unit: Participants] | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis A Antibodies Titre
Time Frame: 6 to 7 months
Population: Received both vaccinations and serum sample at 4 time-points.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Avaxim Pediatric® | Avaxim ® (Adult)
Number analyzed (Participants) | 9 | 7
IU/L
  Baseline (t1) | 9.4 [9.1 to 11] | 9.0 [7.8 to 9.4]
  First dose (t2) | 394.7 [218.65 to 738.4] | 810.6 [317.6 to 2222]
  1 month after (t3) | 343.0 [148.8 to 719.35] | 310.2 [103.45 to 413.45]
  Second dose (t4) | 3975.0 [2282.25 to 21515] | 9372.0 [1676.6 to 17722.5]

ADVERSE EVENTS:
Time Frame: Start of adverse event data collection began when participant first signed consent form. End of adverse event data collection finished 28 days after last dosing.
Arm/Group | Avaxim Pediatric® | Avaxim ® (Adult)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 2/10 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avaxim Pediatric® (N=10) | Avaxim ® (Adult) (N=9)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal Cramping (Gastrointestinal disorders) | 0 | 1
Naseau (General disorders) | 2 | 0
Fever (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT02917577/Prot_SAP_000.pdf